CLINICAL TRIAL: NCT05239364
Title: Ablation of CONseCutive atriaL Tachycardia gUided by Ultra-high-DEnsity Mapping
Brief Title: Ablation of Consecutive Atrial Tachycardia
Acronym: CONCLUDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evangelical Hospital Düsseldorf (Other)
Responsible Party: Principal Investigator, Christian Meyer, Prof. Dr. Christian Meyer, Evangelical Hospital Düsseldorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONCLUDE
Record Dates: First submitted 2022-01-10; First posted 2022-02-14 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Heart Arrhythmia; Heart Diseases; Arrhythmias, Cardiac; Atrial Tachycardia
Keywords: Atrial fibrillation; Atrial tachycardia; Pulmonary vein isolation; Electroanatomical mapping; High density mapping
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Diseases; Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard approach (Experimental): Patients will receive a standard approach for ablation of atrial tachycardia.
  Interventions: Procedure: Catheter ablation
- Minimalized approach (Experimental): Patients will receive a minimalized approach for ablation of atrial tachycardia.
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Catheter-based ablation of arrhythmias using radiofrequency.

SUMMARY:
Ablation of consecutive atrial tachycardia (AT) after ablation of atrial fibrillation (AF) or cardiac surgery can be challenging due to complex substrate and AT mechanisms. A substantial portion of patients is known to show various tachycardias and recurrences occur in a noticeable number of cases. With the availability of novel ultra-high-density mapping techniques characterization and understanding of AT mechanisms and underlying substrate can be improved. Aim of this prospective, multi-center, randomized study is to compare a standard AT ablation approach versus minimalized ablation of the clinical AT in regards to arrhythmia free survival.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive AT subsequent to prior AF ablation procedure or cardiac surgery
* Surface ECG-documentation of AT as primary clinical arrhythmia
* ECG indicating stable, map-able AT (stable activation sequence, and CL stability) with cycle length ≥ 200ms

Exclusion Criteria:

* < 18 years
* No previous atrial fibrillation ablation procedure or cardiac surgery
* Pregnant women or women of childbearing potential without a negative pregnancy test within 48 hours prior to treatment
* History of hemorrhagic diathesis or other coagulopathies
* Contraindications for oral anticoagulation
* Hyper- or hypothyroidism
* Has any condition that would make participation not be in the best interest of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of any sustained arrhythmia (>30 sec.) | 1 year

SECONDARY OUTCOMES:
Inducibility of atrial tachycardia (AT) after ablation of clinical/primary AT (partial success) | Intraprocedural
  Categorical variable (yes/no)
Predictability of secondary AT by analysis of clinical AT map and voltage map | Intraprocedural
Procedure duration time | Intraprocedural
Fluoroscopy time | intraprocedural
Total radiofrequency application time | intraprocedural
Ablated area (cm2) | intraprocedural
Number of blocked lines | intraprocedural
Area of low voltage in sinus map (cm2) | Intraprocedural

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, MD, Principal Investigator — Evangelic Hospital Düsseldorf
Locations (4):
- Germany (4):
  - Evangelic Hospital Düsseldorf, Düsseldorf, North Rhine-Westfalia
  - Evangelic Hospital Hagen-Haspe, Hagen
  - Asklepios St. Georg, Hamburg
  - Universitätsklinikum Schleswig Holstein, Kiel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jungen C, Akbulak R, Kahle AK, Eickholt C, Schaeffer B, Scherschel K, Dinshaw L, Muenkler P, Schleberger R, Nies M, Gunawardene MA, Klatt N, Hartmann J, Merbold L, Jularic M, Willems S, Meyer C. Outcome after tailored catheter ablation of atrial tachycardia using ultra-high-density mapping. J Cardiovasc Electrophysiol. 2020 Oct;31(10):2645-2652. doi: 10.1111/jce.14703. Epub 2020 Aug 11. PMID 32748442
- [Background] Derval N, Takigawa M, Frontera A, Mahida S, Konstantinos V, Denis A, Duchateau J, Pillois X, Yamashita S, Berte B, Thompson N, Hooks D, Pambrun T, Sacher F, Hocini M, Bordachar P, Jais P, Haissaguerre M. Characterization of Complex Atrial Tachycardia in Patients With Previous Atrial Interventions Using High-Resolution Mapping. JACC Clin Electrophysiol. 2020 Jul;6(7):815-826. doi: 10.1016/j.jacep.2020.03.004. Epub 2020 May 27. PMID 32703564
- [Background] Meyer C. High-density mapping-based ablation strategies of cardiac rhythm disorders: the RHYTHMIA experience at new horizons. Europace. 2019 Aug 1;21(Supplement_3):iii7-iii10. doi: 10.1093/europace/euz154. No abstract available. PMID 31400216
- [Background] Takigawa M, Martin CA, Derval N, Denis A, Vlachos K, Kitamura T, Frontera A, Martin R, Cheniti G, Lam A, Bourier F, Thompson N, Wolf M, Massoulie G, Escande W, Andre C, Zeng LJ, Nakatani Y, Roux JR, Duchateau J, Pambrun T, Sacher F, Cochet H, Hocini M, Haissaguerre M, Jais P. Insights from atrial surface activation throughout atrial tachycardia cycle length: A new mapping tool. Heart Rhythm. 2019 Nov;16(11):1652-1660. doi: 10.1016/j.hrthm.2019.04.029. Epub 2019 Apr 18. PMID 31004777